CLINICAL TRIAL: NCT02144883
Title: Telephone Counseling for Pregnant Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Partnership for Smoke-Free Families (PSF) (Unknown)
Responsible Party: Principal Investigator, Shu-Hong Zhu, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB #030310
Record Dates: First submitted 2014-05-15; First posted 2014-05-22 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Smoking
Keywords: telephone counseling
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Materials (Active Comparator): Self-help materials mailed to subjects home.
  Interventions: Behavioral: Self-help materials
- Telephone Counseling and Materials (Experimental): Subjects received up to 9 telephone counseling calls plus self-help quit kit and 5 additional mailings
  Interventions: Behavioral: Telephone counseling; Behavioral: Self-help materials

INTERVENTIONS:
Behavioral: Telephone counseling — Subjects randomized into the telephone counseling condition received one comprehensive pre-quit call lasting about 45 minutes; five follow-up calls during the pregnancy, scheduled according to the risk of relapse after the quit attempt (1, 3, 7, 14, and 30 days after the quit date) one 30-minute pre-birth call scheduled after 36 weeks gestation and two additional follow-up sessions scheduled for 14 and 28 days after the baby's birth. The counseling used a proactive calling procedure in that counselors made all the calls based on agreed-upon dates with the clients. This proactive approach aimed to foster a positive counseling relationship, provide accountability, and create opportunities to address wavering motivation, reduce attrition, and minimize relapse.
  Arms: Telephone Counseling and Materials
Behavioral: Self-help materials — All subjects received a self-help quit kit for pregnant smokers and fact sheets on second-hand smoke and additional tips for quitting while pregnant. Subjects in the counseling intervention group received five additional mailings. These mailings were designed to remind them of their commitment to quitting and of the presence of counseling support if they needed help. Mailings included a pamphlet on pregnancy facts, a refrigerator magnet with the quitline number, and a social support planning worksheet that were sent at 4.5 months, 6 months, and 7.5 months gestation, respectively. They also received a congratulatory card soon after the birth and a brochure with tips for parenting newborns that was sent at one month postpartum.

SUMMARY:
This purpose of the study was to investigate the efficacy of telephone counseling to help pregnant women quit smoking. The investigators tested two hypotheses: 1) telephone counseling increases the overall cessation rate during pregnancy, and 2) the counseling effects can be maintained postpartum.

DETAILED DESCRIPTION:
Smoking during pregnancy increases the risk of low birth weight, premature delivery, fetal and infant death, and children's developmental problems. It is also associated with significant economic costs. Telephone cessation quitlines have been suggested as one good way to reach pregnant smokers.

This randomized controlled trial was embedded into a free statewide telephone cessation quitline in California. The primary component of the intervention was telephone counseling using a structured protocol developed specifically for the pregnant population. The counseling consisted of nine counseling sessions.

A secondary component of the intervention was the mailed materials. Following enrollment in the study all subjects (control and intervention) received a self-help quit kit for pregnant smokers and fact sheets on second-hand smoke and additional tips for quitting while pregnant. Subjects in the counseling intervention group received five additional mailings. These mailings were designed to remind them of their commitment to quitting and of the presence of counseling support if they needed help.

Prior to 36 weeks gestation (in the third trimester), 2-months postpartum, and 6-months postpartum we conducted a brief telephone survey to assess smoking status. The information obtained allowed us to determine 30-day prolonged abstinence rates.

Prior to 36 weeks gestation (in the third trimester), the investigators sent a kit and requested saliva samples be mailed back to biochemically verify smoking status by testing for cotinine and nicotine byproducts.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker willing to quit within one month
* Recent quitters
* First time quitline caller
* Less than 27 weeks gestation
* English and/or Spanish speaking
* Valid phone number
* Valid address
* Gave consent to participate in study and evaluation

Exclusion Criteria:

* Active psychiatric disorder
* Substance or alcohol abuse
* Had been in recovery from alcohol or other substances for less than 6 months
* Planned to use pharmacotherapy
* Insufficient contact information

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1173 (Actual)
Dates: Start 2000-09; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
30 days prolonged abstinence | 6-months postpartum
  Conducted a brief telephone survey to assess smoking status. The information obtained allowed us to determine 30-day prolonged abstinence rates.

SECONDARY OUTCOMES:
Percentage of smokers making a 24-hour quit attempt | <36 weeks gestation
  During evaluation call subjects were asked if they had made a quit attempt that lasted at least 24 hours.
Relapse curve based on quit attempt | Seven months post enrollment
  Kaplan-Meier analysis on the quit attempts over a 6 month period.
Percentage of smokers making a 24-hour quit attempt | 2-months postpartum
  During evaluation call subjects were asked if they had made a quit attempt that lasted at least 24 hours.
Percentage of smokers making a 24-hour quit attempt | 6-months postpartum
  During evaluation call subjects were asked if they had made a quit attempt that lasted at least 24 hours.
7-day cotinine verified abstinence | <36 weeks gestation
  Subjects were asked to submit a saliva sample. This sample was sent to a laboratory to test the cotinine level.
30 days prolonged abstinence | <36 weeks gestation
  Conducted a brief telephone survey to assess smoking status. The information obtained allowed us to determine 30-day prolonged abstinence rates.
  Safety Issue? (FDAAA) No
30 days prolonged abstinence | 2-months postpartum
  Conducted a brief telephone survey to assess smoking status. The information obtained allowed us to determine 30-day prolonged abstinence rates.
  Safety Issue? (FDAAA) No

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Hong Zhu, Ph.D., Principal Investigator — UCSD
Locations (1):
- University of California San Diego California Smokers' Helpline, San Diego, California, United States

REFERENCES:
- [Background] Cummins, S.E., Tedeschi, G.J., Anderson, C.M., Quinlan-Downs, R., Harris, P., Zhu, S.-H. (2007). Telephone counseling for pregnant smokers: essential elements. Journal of Smoking Cessation, 2(2), 36-46.
- [Derived] Cummins SE, Tedeschi GJ, Anderson CM, Zhu SH. Telephone Intervention for Pregnant Smokers: A Randomized Controlled Trial. Am J Prev Med. 2016 Sep;51(3):318-26. doi: 10.1016/j.amepre.2016.02.022. Epub 2016 Apr 4. PMID 27056131